CLINICAL TRIAL: NCT01406353
Title: Early Percutaneous Mitral Intervention Versus Conventional Management in Asymptomatic Moderate Mitral Stenosis
Brief Title: Early Percutaneous Mitral Intervention in Asymptomatic Moderate Mitral Stenosis
Acronym: MITIGATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Duk-Hyun Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0432
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Moderate Mitral Stenosis
Keywords: Mitral Stenosis; Mitral Valvuloplasty
MeSH Terms: conditions — Mitral Valve Stenosis

STUDY DESIGN:
Intervention Model Description: early percutaneous mitral commissurotomy
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Percutaneous Mitral Intervention (Active Comparator): early elective percutaneous mitral commissurotomy within 3 months of enrollment
  Interventions: Procedure: Percutaneous Mitral Commissurotomy
- Conventional Treatment (No Intervention): All patients in the conventional treatment group regularly visit their attending physicians at 3 monthly interval for maintenance of anticoagulation therapy or every year for annual re-evaluation. Patients who become symptomatic during follow-up are referred for percutaneous mitral commissurotomy or mitral valve surgery.

INTERVENTIONS:
Procedure: Percutaneous Mitral Commissurotomy — Percutaneous mitral commissurotomy is performed by experienced interventional cardiologists using the Inoue balloon technique. During the procedure, conventional hemodynamic parameters are monitored. A successful immediate result is defined as a mitral valve area > 1.5 square cm with less than moderate to severe mitral regurgitation.
  Other Names: Percutaneous mitral valvuloplasty
  Arms: Early Percutaneous Mitral Intervention

SUMMARY:
Although percutaneous mitral commissurotomy (PMC) has been accepted as an effective treatment for symptomatic patients with moderate or severe mitral stenosis (MS), most asymptomatic patients are not candidates for PMC owing to the small but inherent procedure-related risks. Asymptomatic patients with MS show good survival rates up to 10 years, but there was a sudden deterioration precipitated by atrial fibrillation or embolism in half of the patients. Because the success rates of PMC were improved to more than 95% in ideal patients from highly selected centers and early PMC may decrease the occurrence of adverse events, such as atrial fibrillation or embolism, experienced centers tend to perform PMC at an early stage of disease. However, the potential benefits of early preemptive PMC in asymptomatic patients should be balanced against the real risks related to the procedure, and further studies of the efficacy of PMC in the prevention of embolism are necessary to extend its indications to asymptomatic patients. To the best of our knowledge, No randomized trials have been performed to ascertain the optimal timing of intervention in asymptomatic patients with significant MS. The early percutaneous MITral Intervention versus conventional manaGement in Asymptomatic moderate miTral stEnosis (MITIGATE) trial was designed to compare clinical outcomes of early intervention with those of a conventional management based on current guidelines in asymptomatic moderate mitral stenosis.

DETAILED DESCRIPTION:
We enroll consecutive asymptomatic patients with moderate mitral stenosis who are candidates for both early percutaneous mitral commissurotomy (PMC) and conventional treatment at 3 centers in Seoul, Korea.

Echocardiographic evaluation is performed before enrollment, immediately after PMC and annually during follow-up. All patients undergo two-dimensional echocardiography and/or transesophageal echocardiography to detect left atrial thrombi. Morphologic features of the mitral valve (MV) are categorized as described previously (14), and total echocardiographic score is obtained by adding the scores for leaflet mobility, thickness, calcification, and subvalvular lesions. The MVA is measured by direct planimetry of the mitral orifice, and MS severity is graded as mild, moderate, or severe when MVA was > 1.5, 1.0 to 1.5, or < 1.0 cm2, respectively. The severity of mitral and tricuspid regurgitation is assessed semiquantitatively or using quantitative methods and classified as mild, moderate, or severe. Pulmonary artery systolic pressure (PAP) is estimated by continuous wave Doppler with the simplified Bernoulli equation.

All study patients regularly visit their attending physicians at 3 monthly interval for maintenance of anticoagulation therapy or every year for annual re-evaluation. Patients in the conventional treatment group who become symptomatic during follow-up are referred for PMC or mitral valve surgery. An embolic event is defined as a systemic embolism fulfilling both prespecified criteria: acute onset of clinical symptoms or signs of embolism and occurrence of new lesions confirmed by imaging studies. A specific diagnosis of cerebral infarction is confirmed by an experienced neurologist and additional brain magnetic resonance imaging is performed if indicated.

We estimate that a sample size of 166 patients would provide 80% power to detect a significant difference with respect to the primary end point at the 2-sided significance level of 0.05, assuming 3-year event rates of 13% in the conventional treatment group and 2% in the early PMC group, and drop-out rate of 5%. These rates are based on the results of our previous study. Analyses are performed on an intention-to-treat basis. To analyze primary outcome, estimates of cumulative event rates are calculated by the Kaplan-Meier method and compared employing the log-rank test. For Kaplan-Meier analysis, we analyze all clinical events by time to first event. Hazard ratios with 95% confidence intervals are derived with the use of the Cox proportional hazards model.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic patients with moderate MS who are potential candidates for early percutaneous mitral commissurotomy

Exclusion Criteria:

* patients with exertional dyspnea
* total echocardiographic score > 10
* moderate to severe mitral regurgitation
* left atrial thrombi
* significant aortic valve disease,
* left ventricle (LV) ejection fraction (EF) <50%
* Doppler-estimated pulmonary artery systolic pressure >50 mmHg
* those who were not candidates for early intervention based on age > 70 years or the presence of coexisting malignancies

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2011-07-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular event | Participants will be followed for the duration of the trial, a minimum follow-up of 10 years
  Composite of cardiovascular mortality, cerebral infarction, systemic embolic events that occurred during follow-up, and PMC-related complications; procedural mortality and urgent MV surgery.

SECONDARY OUTCOMES:
all-cause death and each component of cardiovascular event | Participants will be followed for the duration of the trial, a minimum follow-up of 10 years
  all-cause death and any component of composite primary end point.
Mitral valve replacement | Participants will be followed for the duration of the trial, a minimum follow-up of 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hyun Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University Severance Hospital, Seoul

REFERENCES:
- [Background] Kang DH, Lee CH, Kim DH, Yun SC, Song JM, Lee CW, Song JK, Park SW, Park SJ. Early percutaneous mitral commissurotomy vs. conventional management in asymptomatic moderate mitral stenosis. Eur Heart J. 2012 Jun;33(12):1511-7. doi: 10.1093/eurheartj/ehr495. Epub 2012 Jan 13. PMID 22246444
- [Derived] Kang DH, Park SJ, Lee SA, Lee S, Kim DH, Park DW, Yun SC, Hong GR, Song JM, Hong MK, Park SW, Park SJ. Early percutaneous mitral commissurotomy or conventional management for asymptomatic mitral stenosis: a randomised clinical trial. Heart. 2021 Dec;107(24):1980-1986. doi: 10.1136/heartjnl-2021-319857. Epub 2021 Sep 15. PMID 34526318